CLINICAL TRIAL: NCT05396066
Title: Comparison Between Respiratory and Quadriceps Muscle Fatigability During a Maximal Loading for ICU Weakness Patients
Brief Title: Respiratory and Quadriceps Muscle Fatigability After an ICU Acquired Weakness
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02816-35
Record Dates: First submitted 2022-03-10; First posted 2022-05-31 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: ICU Acquired Weakness
Keywords: ICU acquired weakness; Muscle strength; fatigability; respiratory muscle; Quadriceps muscle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Muscle evaluation — Repeated maximal voluntary contraction

SUMMARY:
Muscle dysfunction can be lead to poor outcomes moreover ICU muscle weakness recovery are not correctly described.

The investigators aimed to assess the ability for quadriceps or respiratory muscles to repeat an effort at a maximal loading.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated at least at 24 Hours
* Maximal inspiratory pressure < 30 centimeter of water
* MRC score < 48/60

Exclusion Criteria:

* Age < 18 years
* Patients with neurological pathology or pre existing neuromuscular dysfunction
* Patient unable to walk 50 meters before ICU admission
* Patient with a thoracic or abdominal surgery
* Inability to carry out maximal voluntary contraction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients weaned from mechanical ventilation and developping ICU muscle weakness diagnosed by a maximal inspiratory pressure and a MRC score
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Respiratory muscle strength | One day
  Respiratory muscle strength will be assessed by Maximal Inspiratory pressure in centimeter of water. The measure will carry out by an electronical manometer
Change in quadriceps muscle strength | One day
  Quadriceps muscle strength will be assessed by Maximal Voluntary contraction of the quadriceps in Newton. The measure will carry out by an electronical dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier du Havre, Montivilliers, Groupe Hospitalier Du Havre, France

REFERENCES:
- [Derived] Machefert M, Prieur G, Aubry S, Combret Y, Medrinal C. Respiratory and limb muscles' ability to repeatedly generate maximal isometric strength in patients with intensive care unit-acquired weakness: an observational study. BMC Anesthesiol. 2025 Mar 20;25(1):134. doi: 10.1186/s12871-025-03008-y. PMID 40114068